CLINICAL TRIAL: NCT01826890
Title: A Randomised Feasibility Study Examining Neurally-adjusted Ventilatory Assist (NAVA) in Patients at High Risk of Prolonged Ventilatory Failure During Recovery From Critical Illness.
Brief Title: Neurally Adjusted Ventilatory Assist in Adults at Risk of Delayed Weaning From Mechanical Ventilation
Acronym: RESTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); King's College London (Other); National Institute for Health Research, United Kingdom (Other Government); JP Moulton Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13/LO/0012
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Adults With Cardiopulmonary Disease at Risk of Prolonged Weaning From Mechanical Ventilation
Keywords: Ventilator Weaning; Mechanical Ventilation; Critical Care; Neurally Adjusted Ventilatory Assist; Diaphragm
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAVA technology (Experimental): Following randomisation, a NAVA catheter will be introduced. The Electrical Activity of the Diaphragm (EAdi) will be viewed primarily to ensure a minimum level of diaphragm activation during the weaning phase. NAVA mode suitability/safety assessments will be conducted in all patients prior to the first initiation of the NAVA mode. The NAVA preview function on the Maquet Servo-i ventilators will be used to transfer from the previous mode to the NAVA mode, and the assessment will last for a maximum of 30 minutes. We are recommending the use of the NAVA ventilation mode during the weaning period. Following the commencement of weaning, sedation holds and spontaneous breathing trials will be conducted according to local protocols.
  Interventions: Other: NAVA Technology
- Standard Care (No Intervention): A NAVA catheter will be inserted following randomisation. The NAVA capabilities of the ventilator will be disabled. Patients will be ventilated according to local weaning protocol as per current standard care with either Pressure Support, Synchronised Intermittent Mandatory Ventilation, Volume Controlled Ventilation, Pressure Controlled Ventilation or Pressure Regulated Volume Controlled Ventilation. Following the commencement of weaning, sedation holds and spontaneous breathing trials will be conducted according to local protocols.

INTERVENTIONS:
Other: NAVA Technology — Use of NAVA technology: Diaphragmatic monitoring and NAVA ventilation mode
  Other Names: Neurally Adjusted Ventilatory Assist; NAVA
  Arms: NAVA technology

SUMMARY:
Many patients admitted to intensive care have heart or lung problems. Patients with these conditions often require longer durations of support from breathing machines. Survival and long-term recovery are improved if the investigators can remove the breathing support quickly. In this study, the investigators will focus on patients with severe lung or heart disease to examine whether a particular type of breathing machine (NAVA ventilator) will allow us to remove breathing support more quickly and with less need for sedative medications, when compared to current practice.

DETAILED DESCRIPTION:
In this study, we will compare the use of Neurally Adjusted Ventilatory Assist technology (the NAVA ventilation mode and the monitoring capabilities) against standard care in patients who are at risk of prolonged periods of mechanical ventilation.

Study aim

To inform the design of a definitive randomised controlled trial (RCT) by undertaking feasibility testing, evaluation of the proposed NAVA intervention and evaluation of the proposed outcomes.

Feasibility outcomes

* Number of eligible patients
* Assessment of screening and recruitment methods
* The willingness of clinicians to allow recruitment
* The willingness of participants to be randomised
* Assessment of the randomisation process
* Staff attitudes and training needs
* Protocol compliance (barriers to the use of NAVA ventilation)

Intended primary outcomes of the main study

*Ventilator-free days (day 28)

There are a number of secondary outcomes that include:

* Total sedation / hypnotic / analgesic dose
* Ventilator free days (day 90)
* Duration of invasive mechanical ventilation (MV)
* Duration of MV (including Non-invasive ventilation (NIV))
* Duration of post extubation NIV
* Incidence of delirium (CAM-ICU)
* Change in sequential organ failure assessment (SOFA) score from baseline to day 3, 7, 14 and 28
* ICU and hospital length of stay
* Day 28, ICU discharge, hospital discharge and 90 day post randomisation survival
* Agitation / comfort (Richmond Agitation and Sedation Score (RASS) plus Visual *Analogue Scale where possible)
* Frequency of sedation / analgesic / hypnotic bolus doses
* Ventilator associated pneumonia (developed 48 hours after study entry)
* Unplanned device removal (eg. ET tubes, catheters etc.)
* Patient-ventilator asynchrony
* Duration in each ventilation mode
* Change in the electrical activity of the diaphragm (EAdi)
* Health Resource Group costs
* Quality of life at 90 days - SF36 questionnaire

STUDY DESIGN

A pilot feasibility, single centre, open label randomised controlled study. In summary, group one will receive standard care and group two will receive standard care with the addition of NAVA technology.

POPULATION

Intubated, critically ill or high-risk elective peri-operative adult patients who are at greatest risk of difficult or prolonged weaning: those with pre-existing cardiopulmonary dysfunction.

Inclusions

ICU admissions who are likely to remain intubated and ventilated for greater than 48 hours with a diagnosis of one or a combination of:

1. COPD
2. Left and/or right ventricular heart failure
3. Mild, moderate or severe (Berlin criteria) Acute Respiratory Distress Syndrome (ARDS)

All diagnoses must be documented in the medical notes. There must be evidence of a specialist consultant diagnosis, or a non-specialist doctor diagnosis with either objective test results (spirometry, CT, lung biopsy, cardiac echo) and/or prescribed treatment.

Exclusions

* Less than 18 years old or pregnant.
* Inability to conduct protocol (e.g. research staff or NAVA technology unavailable).
* No personal or nominated consultee available or assent declined.
* Greater than 96 hours from intubation.
* Greater than 24 hours in the weaning phase.
* Patient likely to die/have treatment withdrawal within 48 hours.
* Contraindication to passing NG tube.
* Patients with primary neurological cause of ventilator dependence.
* High spinal injury above C6; severe traumatic brain injury (Glasgow Coma Score < 8).
* Suspected or proven hypoxic brain injury.
* Physician refusal / physician wishes to use NAVA.
* Hepatic encephalopathy greater than grade one.
* Domiciliary ventilation (except Continuous Positive Pressure (CPAP)or Bi-level Positive Airway Pressure (BIPAP) used for sleep disordered breathing).
* Enrollment in another interventional clinical trial in the last 30 days.
* Non-English speakers where inadequate translation available to allow informed consent.

STUDY SITE

Three adult ICUs at KCH NHS Foundation Trust, London.

SAMPLE SIZE

76 patients will be recruited to estimate an anticipated compliance of 75% (95% confidence interval of +/- 10%).

FOLLOW-UP SF-36 will occur at 90 days post ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

ICU admissions who are likely to remain intubated and ventilated for greater than 48 hours with a diagnosis of one or a combination of:

1. COPD
2. Left and/or right ventricular heart failure
3. Mild, moderate or severe (Berlin criteria) Acute Respiratory Distress Syndrome (ARDS)

All diagnoses must be documented in the medical notes. There must be evidence of a specialist consultant diagnosis, or a non-specialist doctor diagnosis with either objective test results (spirometry, CT, lung biopsy, cardiac echo) and/or prescribed treatment.

Exclusion Criteria:

* Less than 18 years old or pregnant
* Inability to conduct protocol (e.g. research staff or NAVA technology unavailable)
* No personal or nominated consultee available or assent declined
* Greater than 96 hours from intubation
* Greater than 24 hours in the weaning phase
* Patient likely to die/have treatment withdrawal within 48 hours
* Contraindication to passing NG tube
* Patients with primary neurological cause of ventilator dependence
* High spinal injury above C6; severe traumatic brain injury (Glasgow Coma Score < 8)
* Suspected or proven hypoxic brain injury
* Physician refusal / physician wishes to use NAVA
* Hepatic encephalopathy greater than grade one
* Domiciliary ventilation (except CPAP/BIPAP used for sleep disordered breathing)
* Enrollment in another interventional clinical trial in the last 30 days
* Non-English speakers where inadequate translation available to allow informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-05; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Protocol compliance | 28 days
  Total time in the NAVA ventilation mode as a proportion of total time in an assisted spontaneous weaning ventilation mode within 28 days from randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Hadfield, Principal Investigator — King's College Hospital NHS Trust; Phillip A Hopkins, Study Chair — King's College Hopspital NHS Foundation Trust; Nicholas Hart, Study Director — Guy's and St Thomas' NHS Foundation Trust; Gerrard F Rafferty, Study Director — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Hadfield DJ, Rose L, Reid F, Cornelius V, Hart N, Finney C, Penhaligon B, Molai J, Harris C, Saha S, Noble H, Clarey E, Thompson L, Smith J, Johnson L, Hopkins PA, Rafferty GF. Neurally adjusted ventilatory assist versus pressure support ventilation: a randomized controlled feasibility trial performed in patients at risk of prolonged mechanical ventilation. Crit Care. 2020 May 14;24(1):220. doi: 10.1186/s13054-020-02923-5. PMID 32408883